CLINICAL TRIAL: NCT04821895
Title: A Taiwanese Oncogenetic Panel and Integrated Clinical Data Registration Study for Wild Type Gastrointestinal Stromal Tumor Patients (TOPICS-GIST)
Brief Title: Oncogenetic Panel and Integrated Clinical Data Registry Study for Wild Type Gastrointestinal Stromal Tumor Patients
Acronym: GIST
Status: Active, not recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Tri-Service General Hospital (Other); Mackay Memorial Hospital (Other); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); Taichung Veterans General Hospital (Other); Changhua Christian Hospital (Other); Kaohsiung Veterans General Hospital. (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T1221
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
Keywords: Gastrointestinal Stromal Tumor(GIST); Oncogenetic Panel
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Biospecimen Retention: Samples Without DNA — oncopaenl test
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The genetic background for cancer treatment may also be different among different areas and races. There is lack of Taiwanese data of genetic alterations in cancer patients. To understand the landscape of genetic aberrations of cancer in Taiwan, large scale survey of the cancer patients is indicated. In this pilot study, the investigators want to evaluate the landscape of genetic aberrations in cancer patients via oncopaenl test and collect the clinical data of the patients. The result of the oncopanel test will be returned to patient and their attending physician for reference of their further treatment. In addition, the investigators want to correlate the clinical outcome with the genetic aberrations of the cancer patients in Taiwan. Gastrointestinal stromal tumor (GIST) is a rare cancer compared with the other solid tumors. C-KIT or PDGFRA mutation is found in approximately 85-90% of GISTs. Imatinib, a tyrosine kinase inhibitor targeting c-KIT, has been used to treat advanced GIST successfully since 2000. However, resistance to imatinib may develop either via secondary mutation of c-KIT or primary resistance to those with wild type c-KIT and PDGFRA. Although sunitinib and regorafenib have been approved as second and third line of treatment for advanced GIST, the progression free survival were only 6.8 and 4.8 months, respectively. The genetic landscape of GIST with wild type c-KIT and PDGFRA was less studied. In the current study, the investigators want to focus on the GISTs with wild type c-KIT and PDGFRA to perform the NGS oncopanel for these patients. Then the investigators can understand the genetic aberrations of these patients (wild type GIST) and help for searching the potential treatment targets to them.

DETAILED DESCRIPTION:
Cancer is the most common cause of death in Taiwan since 1982. The incidence of cancer is increasing worldwide, including Taiwan. Cancers in early stage can usually treated with surgery with a good prognosis. However, the prognosis for recurrent, locally advanced or metastatic cancers are poor with a shorter survival. Systemic treatments are usually indicated for these patients. Chemotherapy is the main stay for advanced cancer patients. However, the advances in the understanding of cancer biology and identification of targeted therapeutics not only increase the treatment strategies of cancer but also improves the survival and quality of life of the cancer patients. There are more and more molecularly targeted therapy developed and approved for the treatment of advanced cancer patients currently, which makes the beginning of precision cancer medicine. There are more and more treatments can be used based on the genetic aberrations of the cancers. Because one cancer type may habor various genetic aberrations, it is not enough to check only one or a few genes for a patient to choose the adequate treatment. Because the advance in multiplex genomic test, several NGS-based cancer-associated genetic panel test (oncopanel) have been developed and used to identify the genetic alterations in each patient, particularly the actionable genes. Large scale checks of oncopanel have been executed in US. The study showed the genetic alterations in various cancer types and 11% of the patients had further molecular targeted therapy based on the result of the oncopanel test. The similar program was done in Japan. Moreover, the oncopanel test have been implicated in their clinical practice and the cost was reimbursed by the government in Japan and Korea recently. The precision medicine and such personalized treatment is the trend for cancer treatment. The trend of such treatment patterns is also observed in Taiwan. The genetic background for cancer treatment may also be different among different areas and races. There is lack of Taiwanese data of genetic alterations in cancer patients. To understand the landscape of genetic aberrations of cancer in Taiwan, large scale survey of the cancer patients is indicated. In this pilot study, the investigators want to evaluate the landscape of genetic aberrations in cancer patients via oncopaenl test and collect the clinical data of the patients. The result of the oncopanel test will be returned to patient and their attending physician for reference of their further treatment. In addition, the investigators want to correlate the clinical outcome with the genetic aberrations of the cancer patients in Taiwan. Gastrointestinal stromal tumor (GIST) is a rare cancer compared with the other solid tumors. C-KIT or PDGFRA mutation is found in approximately 85-90% of GISTs. Imatinib, a tyrosine kinase inhibitor targeting c-KIT, has been used to treat advanced GIST successfully since 2000. However, resistance to imatinib may develop either via secondary mutation of c-KIT or primary resistance to those with wild type c-KIT and PDGFRA. Although sunitinib and regorafenib have been approved as second and third line of treatment for advanced GIST, the progression free survival were only 6.8 and 4.8 months, respectively. The genetic landscape of GIST with wild type c-KIT and PDGFRA was less studied. In the current study, wthe investigators want to focus on the GISTs with wild type c-KIT and PDGFRA to perform the NGS oncopanel for these patients. Then the investigators can understand the genetic aberrations of these patients (wild type GIST) and help for searching the potential treatment targets to the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed GIST.
2. The tumors can be resected, unresectable, recurrent or metastatic and the patients had ever received, are receiving or will receive systemic treatment (adjuvant, neoadjuvant or salvage TKI or other targeted agents)
3. The tumors were tested for wild type c-KIT and PDGFRA.
4. There are archived tumor samples available or the patients agree to do tumor biopsy for oncopanel test if there is no tumor sample or not enough tumor sample available.
5. The patients who are systemic treatment naïve or have received prior systemic treatment are all eligible.
6. Age - the legal age.
7. Life expectancy greater than 6 months
8. Capable of understanding and complying with the protocol requirements and signed informed consent.

Exclusion Criteria:

* Patients will be excluded from the study if they meet any of the following criteria:

  1. Inability and unwillingness to give informed consent
  2. Patients do not agree to provide archived tumor samples and blood samples or they do not agree to do tumor biopsy when archived tumor samples are not available.
  3. Patients refused for collection of clinical data and follow up.
  4. Mental status is not fit for further treatment or data collection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wild Type Gastrointestinal stromal tumor (GIST)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-28 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
genetic profiles in gastrointestinal stromal tumor (GIST) patients | 5-year time frame
  To evaluate the genetic profiles in gastrointestinal stromal tumor (GIST) patients without c-KIT and PDGFRA mutation (wild type) in Taiwan.

SECONDARY OUTCOMES:
Collect clinical data of wild type GIST patients | 5-year time frame
  Collect clinical data of wild type GIST patients
To correlate the clinical characteristics, treatment and outcome of wild type GIST patients with the genetic profile in Taiwan. | 5-year time frame
  To correlate the clinical characteristics, treatment and outcome of wild type GIST patients
To help for search the potential targeted agents for the treatment of these wild type GIST patients | 5-year time frame
  To help for search the potential targeted agents for the treatment of these wild type GIST patients

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Jen Tsai, M.D., Principal Investigator — National Health Research Institutes, Taiwan; Li-Tzong Chen, Ph.D, Study Chair — leochen@nhri.org.tw
Locations (11):
- Taiwan (11):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided